CLINICAL TRIAL: NCT02947477
Title: EmoTrak, Ecological Momentary Assessment of Emotion, Stress and Satisfaction Among Residents
Brief Title: Emotion Tracking Study for Residents
Acronym: ETSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RAPFUNDEKMAN
Record Dates: First submitted 2016-10-24; First posted 2016-10-28 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Stress, Emotional
MeSH Terms: conditions — Stress, Psychological

ARMS (2):
- Treatment (Experimental): The EMA intervention uses twice-a-day interactive questions for emotion tracking including type of emotion, intensity of emotion, trigger to emotion and response to emotion through an Iphone app designed for the study. The study users receive individualized feedback about their daily reporting of emotions, sleep and stress.The study tracking is for 14 days.
  Interventions: Behavioral: EmoTrak
- Control (No Intervention): The control arm does nothing for 14 days and then receives the 14 day emotion tracking listed above.

INTERVENTIONS:
Behavioral: EmoTrak — Ecological Momentary Assessment of Emotion through Iphone App
  Arms: Treatment

SUMMARY:
The proposed study will develop and pilot a fourteen-day assessment tailored for the high-demand schedule of residents through a smart phone intervention, EmoTrak.EmoTrak uses ecological measurement assessment (EMA), which solicits real-time user feedback at various time points across a series of days or weeks.

DETAILED DESCRIPTION:
The investigators will perform a randomized controlled trial that compares residents, using EmoTrak with a wait list control group. After two weeks, the active control group becomes the treatment group. All participants will be evaluated four times from at baseline to two months. The measures to explore for any pre and post change are stress reduction on the emotional exhaustion scale of the Maslach Burnout Inventory (MBI) and improved resilience on the Perceived Stress Scale (PSS).

ELIGIBILITY:
Inclusion Criteria:

* Currently in Residency or Fellowship at UCSF

Exclusion Criteria:

* Not having an Iphone

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12-17 (Actual); Study Completion 2017-12-17 (Actual)

PRIMARY OUTCOMES:
Retention of Participants Iphone App for Residents | 14 days
  Quantify amount of drop out through out the 14 day study and how many reports are responded two daily
Acceptability of Iphone App for Residents Online Evaluation and Mini Interviews | 30 days
  Evaluate online questions and qualitative mini interviews about the usability of the app

SECONDARY OUTCOMES:
Real Time Assessment Comparison to Standardized Measures | 35 days
  Compare Pre, Post and Midway Assessments of Stress, Burnout and Emotion Awareness with daily, longitudinal measures to explore relationships between these sources of data.
Ecological Assessment of Emotions Compared to Standardized Emotion Awareness Measures, PANAS | 14 days
  Comparing the daily reports of emotions in comparison to the PANAS scale of last week of experienced emotions
Ecological Assessment of Stress Compared to Standardized Perceived Stress and Emotional Exhaustion from the Maslach Burnout Inventory | 14 days
  Comparing the daily reports of stress s in comparison to the week of stress as measured by PSS and MBI.

OTHER OUTCOMES:
Exploratory Analysis of Reduction in Pre and Post Reported Emotional Exhaustion on the MBI | 30 days
  Exploratory analysis of pre and post reduction of participants using EmoTrak versus wait list control on Emotional Exhaustion subscale of Burnout.
Exploratory Analysis of Reduction in Pre and Post Reported Stress on PSS and MBI | 30 days
  Exploratory analysis of pre and post improvements of participants using EmoTrak versus wait list control on Perceived Stress.
Exploratory Analysis of Increase in Pre and Post Reported Resilience on the CDRisc | 30 days
  Exploratory analysis of pre and post improvements of participants using EmoTrak versus wait list control on a measure of resilience to dealing with stress.

CONTACTS AND LOCATIONS:
Overall Officials: Eve Ekman, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riess H, Kelley JM, Bailey RW, Dunn EJ, Phillips M. Empathy training for resident physicians: a randomized controlled trial of a neuroscience-informed curriculum. J Gen Intern Med. 2012 Oct;27(10):1280-6. doi: 10.1007/s11606-012-2063-z. Epub 2012 May 2. PMID 22549298